CLINICAL TRIAL: NCT06708637
Title: An Open-Label, Multi-Center, Single-Arm Study to Evaluate the Ocular Safety and Usability of FYB203 Pre-filled Syringe (PFS)
Brief Title: Ocular Safety and Usability Study for FYB203 PFS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Formycon AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FYB203-04-01
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Age-Related Macular Degeneration; Branch Retinal Vein Occlusion with Macular Edema; Central Retinal Vein Occlusion with Macular Edema; Diabetic Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FYB203 2 mg (0.05 mL of 40 mg/mL) (Experimental): FYB203 provided in a pre-filled syringe (PFS), containing 2 mg of 40 mg/mL aflibercept in 0.05 mL for intravitreal (IVT) administration
  Interventions: Drug: FYB203 2 mg (0.05 mL of 40 mg/mL)

INTERVENTIONS:
Drug: FYB203 2 mg (0.05 mL of 40 mg/mL) — IVT administration of FYB203 in a PFS
  Other Names: aflibercept-mrbb

SUMMARY:
The objective of the study is to assess the ocular safety of the FYB203 pre-filled syringe in terms of preparation and administration by Retina Specialists in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Study eye deemed to be indicated for aflibercept IVT injection therapy at the discretion of the Investigator.
2. Written and signed informed consent form (ICF) obtained before any study-related procedures.
3. Had a confirmed diagnosis in one or both eyes of neovascular (wet) AMD or macular edema following RVO or DME or DR.
4. Qualified for treatment with aflibercept according to the United States Prescribing Information.
5. Aged ≥18 years at the time of signing ICF.
6. If a subject was already on an aflibercept regimen, timing of study participation was correlated with the regimen.
7. Male study subject (if his female spouse/partner was of childbearing potential) must have confirmed that he was using two acceptable methods for contraception (one of which must be a barrier method) starting at signing ICF and throughout the clinical study period and for 3 months after IP administration. Male study subject must have agreed to inform his partner of participation in the study and the need to avoid pregnancy. Surgically sterilized and non sexually active male subjects did not require any additional use of contraception.
8. Male study subject agreed not to donate sperm starting from screening and throughout the clinical study period and for 3 months after IP administration.
9. Female study subject was categorized by at least one of the following:

   * Not a woman of childbearing potential as described in Appendix 3 of the study protocol prior to signing ICF, or
   * Surgically sterile or had undergone a hysterectomy as categorized in Appendix 3 of the study protocol at least 1 month prior to signing ICF, or
   * Was using a highly effective contraception. All females of childbearing potential were required to use highly effective contraception (as described in Appendix 3 of the study protocol) starting at signing ICF and throughout the clinical study period and for 3 months after IP administration.
10. Female study subject must not be lactating and must not be breastfeeding at screening until 3 months after IP administration.
11. Female study subject must not donate ova starting at signing ICF and throughout the clinical study period and for 3 months after IP administration.

Exclusion Criteria:

1. Had received IVT injection in the study eye within 3 months prior to Day 1 with any anti vascular endothelial growth factor therapy other than aflibercept products (ege.g., Eylea).
2. Intraocular corticosteroid administration in the study eye within 30 days prior to Day 1.
3. Had fever or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non cutaneous) infection within 1 week prior to Day 1.
4. History or evidence of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection in the last month prior to signing ICF or had been in confirmed contact with SARS-CoV-2 positive subjects in the last 2 weeks before dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence and occurrence of ocular and non-ocular Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring after IVT injection | 2 days
  To assess the ocular safety of the FYB203 PFS in terms of preparation and administration by Retina Specialists.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Campbell, California
  - Research Site, Long Beach, California
  - Research Site, Redlands, California
  - Research Site, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No